CLINICAL TRIAL: NCT00002876
Title: A PHASE II TRIAL OF ETOPOSIDE AND CISPLATIN IN THE TREATMENT OF RECURRENT EPENDYMOMAS
Brief Title: Etoposide Plus Cisplatin in Treating Patients With Recurrent Ependymomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Randolph S. Marks, MD, Mayo Clinic
Purpose: Treatment
Other Study IDs: CDR0000065162; P30CA015083 (NIH); 907253 (Other: Mayo Clinic Cancer Center); V96-1072 (Other: NCI Protocol); 394-91 (Other: Mayo Clinic IRB)
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult myxopapillary ependymoma; adult anaplastic ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Ependymoma | interventions — Cisplatin; Etoposide

INTERVENTIONS:
Drug: cisplatin
Drug: etoposide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients with recurrent ependymomas following radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the efficacy and toxicity of etoposide and cisplatin in patients with recurrent ependymomas.

OUTLINE: All patients receive cisplatin followed by etoposide on days 1-3. Treatment repeats every 4 weeks for a total of 6 courses unless disease progression or unacceptable toxicity intervenes. The etoposide dose may be increased by 10% on subsequent courses if the white blood cell and platelet nadirs on the previous course are at least 3,000 and 100,000, respectively. Patients are followed every 2 months for 6 months, then every 3 months for 4.5 years.

PROJECTED ACCRUAL: A total of 35 patients will be entered over approximately 7 years if there are 3-8 responses in the first 13 patients and 7-9 responses in the first 25 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed ependymoma that is recurrent after radiotherapy Histologic confirmation of recurrence encouraged but not required in patients with pure ependymoma at diagnosis and unequivocal radiologic evidence of recurrence Histologic confirmation of recurrence required in patients with mixed histology at diagnosis Ependymoma at least 80% of histology No subependymoma Measurable or evaluable disease on imaging exam

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-3 Hematopoietic: WBC at least 3,500 Platelets at least 130,000 Hepatic: Bilirubin no greater than 0.3 mg/dL above normal Renal: Creatinine no greater than 0.3 mg/dL above normal Cardiovascular: No NYHA class III/IV status Other: No uncontrolled infection No pregnant or nursing women Negative pregnancy test required of fertile women Effective contraception required of fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior cisplatin or etoposide At least 4 weeks since chemotherapy (6 weeks since nitrosoureas) Endocrine therapy: Steroid dose stable for at least 1 week prior to entry if indicator lesion in CNS Radiotherapy: See Disease Characteristics At least 4 weeks since radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 1991-10; Primary Completion 1998-04 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randolph S. Marks, MD, Study Chair — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota